CLINICAL TRIAL: NCT05787288
Title: Clinical Study on the Safety and Efficacy of Mesenchymal Stem Cell Exosomes in the Treatment of Coronavirus Infection.
Brief Title: A Clinical Study on Safety and Effectiveness of Mesenchymal Stem Cell Exosomes for the Treatment of COVID-19.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: REGEN-αGEEK (SHENZHEN) MEDICAL TECHNOLOGY CO., LTD. (Unknown)
Responsible Party: Principal Investigator, Xiaoying Huang, Vice President of First Affiliated Hospital of Wenzhou Medical University, First Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2022-205
Record Dates: First submitted 2023-03-27; First posted 2023-03-28 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19, Exosomes, Mesenchymal Stem Cell
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Nebulized Mesenchymal Stem Cell Exosomes-derived extracellular vesicles twice a day (BID) for 5 days
  Interventions: Biological: Extracellular Vesicles from Mesenchymal Stem Cells
- Control Group (Sham Comparator): Nebulized saline solution twice a day (BID) for 5 days
  Interventions: Biological: Extracellular Vesicles from Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Extracellular Vesicles from Mesenchymal Stem Cells — Umbilical cord mesenchymal stem cell-derived extracellular vesicle preparation; Specification: 5ml, with extracellular vesicle concentration of 1 × 109 particles/ml in the preparation;

SUMMARY:
This clinical study aims to investigate the safety and efficacy of nebulized inhalation of extracellular vesicles derived from mesenchymal stem cells combined with standard therapy for COVID-19-infected individuals. The primary objective is to determine whether nebulized MSC-secreted extracellular vesicles may be a feasible approach to alleviate COVID-19-induced lung injuries and promote recovery. Participants will be allocated to receive either nebulized MSC-secreted extracellular vesicles twice a day (BID) for 5 days as the test group or nebulized saline solution twice a day for 5 days as the control group. Researchers will compare the test and control groups to evaluate the safety and efficacy of extracellular vesicles in combination with standard therapy.

DETAILED DESCRIPTION:
1. Background 1.1. New Coronavirus Infection and Current Medical Strategies The 2019 coronavirus disease (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has been raging for over three years, causing more than 5 million deaths worldwide. The World Health Organization has declared COVID-19 pneumonia a global pandemic and a public health emergency[1]. Although diagnostic efficiency and treatment accuracy have improved, the overall treatment effect is still limited. The main causes of death include severe pneumonia, acute respiratory distress syndrome (ARDS), pulmonary edema, or multiple organ failure[2]. Among them, ARDS is the most severe. Pathological studies have shown that the pathogenesis of ARDS is mainly due to the immune response induced by the coronavirus attacking alveolar cells; immune cell infiltration leads to destruction of the pulmonary capillary endothelial structure, causing plasma, plasma proteins, and blood cells to enter the lung interstitium and alveolar cavity, forming pulmonary edema. Due to the destruction of the alveolar epithelial tissue, a large amount of edema fluid enters the alveoli, resulting in limited diffusion function of the alveoli and inability to perform normal respiratory function. At the same time, with the aggravation of tissue damage, cells further release various inflammatory factors to form a so-called cytokine storm, which finally completely destroys most of the pulmonary alveoli and bronchial respiratory structures, causing severe ventilation-perfusion imbalance and ultimately death of the patient[3].

   In this global emergency event of coronavirus, the main medical strategy to combat COVID-19 is to use antibiotics and antiviral drugs to block the virus replication cycle and suppress host inflammation. This strategy has led to effective supportive and symptomatic treatment in some cases, even yielding promising results, but it is not the ultimate treatment for this infection. For example, immune regulation interventions like tocilizumab (IL-6 receptor blocker), adalimumab (anti-TNF antibody), and eculizumab (anti-C5 antibody) can effectively relieve patient symptoms but cannot cure the disease fundamentally. In fact, there are two major characteristics of COVID-19 pneumonia: first, people with low immunity are more susceptible to COVID-19[4], and second, the main target organ is the lungs[5]. In fact, respiratory failure has been reported as one of the main causes of death from COVID-19[6], and autopsies have shown lung damage, significant exudative reactions, and pulmonary embolism in many patients[7].

   1.2. Mesenchymal Stem Cell Exosomes Mesenchymal stem cells (MSCs) have been shown to have comprehensive and powerful immunomodulatory and regenerative functions[8]. MSCs can combat cell death associated with the pathogenesis of chronic obstructive pulmonary disease (COPD), idiopathic pulmonary fibrosis, asthma, ARDS, and pulmonary hypertension, and promote cell regeneration[9,10]. Exosomes are one of the key paracrine effectors secreted by MSCs and are considered attractive candidates for alternative MSC therapy due to their biocompatibility similar to parent cells and their ability to maintain healing properties[11]. Under physiological and pathological conditions, exosomes play a key role in intercellular communication by transporting various biomolecules such as miRNA and proteins to target cells[12]. Unlike apoptotic bodies and microvesicles derived from the cell surface, exosomes are produced through the endocytic pathway and load cytoplasmic content of the parent cell. Therefore, they are mini versions of parent cells, mimicking some of their physiological characteristics. Compared to cell counterparts, the non-toxicity, low immunogenicity, high stability, ease of storage, and potential for mass production as ready-made products are several advantages of exosomes, which have led to their expansion in clinical applications as new therapeutic alternatives. In addition, the natural function of exosomes allows them to deliver their membrane and cytoplasmic bioactive components from parent cells to target cells through membrane fusion[13]. There are also other unique characteristics, including the natural ability to cross biological barriers such as the blood-brain barrier (BBB). Furthermore, biocompatibility is another characteristic. Due to their origin from biological sources and inherent targeting ability, exosomes have been used as carriers of drug components in preclinical studies[14].

   1.3. Mechanism of Mesenchymal Stem Cell-derived Exosomes Treatment MSC-derived exosomes inherit immune suppressive properties from their parent cells, and MSC-evs may use various mechanisms to balance the immune system's function. One key mechanism is reprogramming and altering the phenotype of various immune cells. For example, the ability of MSC-derived exosomes to promote the survival of alveolar macrophages and shift their phenotype from pro-inflammatory (M1) polarization to anti-inflammatory (M2) polarization has been demonstrated in at least two studies. These findings suggest that exosomes can serve as viable alternatives to their parent cells, and this ability has also been reported to alter the Treg/Teff ratio to increase Treg and promote the secretion of anti-inflammatory cytokines[15,16].

   In multiple models, MSC-evs have similar therapeutic characteristics to MSCs, are easier to prepare, store and transport to the bedside, and avoid some limitations of cell therapy, such as the risk of pulmonary embolism and tumor formation. In recent years, MSC-evs have received widespread attention as biomarkers of pathogenesis and therapeutic drugs for a variety of diseases. In addition, MSC-secreted exosomes can regulate immunity through interaction with immune cells and inhibit inflammatory responses through cytokines[17,18]. Numerous studies have shown that MSC-secreted exosomes can be used to treat immune deficiencies, inflammation, ARDS, and other pulmonary diseases[19,20], so MSC-secreted exosomes may also be effective in treating the lung inflammation caused by COVID-19.Exosomes are one of the main active ingredients secreted by stem cells and are 30-150 nm in size. After nebulization, exosomes can directly reach the bronchioles and alveoli, which is conducive to the maximum absorption of drugs[21]. Multiple clinical trials have shown that intravenous infusion of MSCs and MSC-evs for the treatment of severe lung damage caused by SARS-CoV-2 is safe and effective[22], and in the case of lung injury, the nebulization route provides a particularly effective drug delivery method to target lung sites. Therefore, we speculate that nebulized MSC-secreted exosomes may be an effective method for reducing COVID-19 lung damage and promoting recovery.

   1.4. Clinical Case Studies of Stem Cell-derived Exosomes Recently, the inhaled anti-COVID-19 drug Exo-CD24, led by Israeli medical center expert Nadir Arber, which is a combination of exosomes and CD24 protein, has shown promising results in early clinical trials. The drug was able to cure 29 out of 30 severe patients within 5 days of treatment and has the potential to treat COVID-19 patients within 3-5 days. Although Exo-CD24 has not yet passed phase III testing, it has shown great potential in the future[23]. The US FDA has approved the use of extracellular vesicles (EVS) for the treatment of COVID-19 through a Phase I/II trial conducted by Direct Biologics. ExoFlo, the EVS used, restores the health and vitality of patients by reducing sustained inflammation, promoting the revascularization of damaged tissue, and reshaping scar tissue. Domestic clinical studies have also been initiated, clinical research at the Fifth People's Hospital of Wuxi City, Jiangsu Province has confirmed that nebulized umbilical cord mesenchymal stem cell-derived extracellular vesicles are a safe and viable treatment for COVID-19. The study was published in Stem Cell Reviews and Reports in June of this year and included seven patients diagnosed with COVID-19 pneumonia, including two severe cases (Patients 2 and 4) and five mild cases (Patients 1, 3, 5, 6, and 7). No acute allergic reactions such as throat or tongue swelling, rash, shortness of breath, dizziness, vomiting, or hypotension were observed in any of the patients within two hours after nebulization treatment. There were also no reported adverse events or secondary allergic reactions following treatment. Chest CT scans showed a decrease in lung lobe nodule density and absorption of lung lesions in both severe and mild patients after nebulized treatment with MSC-derived extracellular vesicles[21]. Joint research by Ruijin Hospital and Jinyintan Hospital is being conducted on nebulized COVID-19 treatment using adipose-derived human allogeneic mesenchymal stem cell-derived exosomes (HAMSCs-Exos). Seven critically ill COVID-19 patients were treated with HAMSC-Exos via nebulization inhalation, and all patients tolerated the treatment well without evidence of adverse events or clinical instability during or immediately after nebulization. All patients showed an increase in serum lymphocyte count (median of 1.61×10^9/L vs 1.78×10^9/L), and lung lesions were reduced to varying degrees in all patients after inhaling HAMSC-Exos aerosols, with four patients showing significant improvement. Preliminary results suggest that participants' lung injuries were significantly improved[21].

   However, most clinical trials using stem cell exosomes for COVID-19 infection have the following issues: (a) small sample size, making it difficult to effectively demonstrate the advantages of stem cell exosomes in COVID-19 treatment; (b) lack of a control group; (c) use of traditional two-dimensional production methods, making it difficult to scale up production of large quantities of exosomes for clinical treatment; and (d) lack of in-depth mechanism exploration for relevant phenomena. These problems hinder progress in the use of stem cell exosomes for COVID-19 infection treatment. To address these issues, this project proposes combining nebulized umbilical cord mesenchymal stem cell exosomes with conventional treatment to treat middle to severe COVID-19 patients and evaluate its safety and efficacy.
2. Research Objective This study aims to evaluate the safety and effectiveness of umbilical cord mesenchymal stem cell-derived exosomes (nebulized) combined with conventional therapy for the treatment of moderate, severe, and critically ill COVID-19 patients through a multicenter, randomized controlled, single-blind clinical trial.
3. Research Design This study adopts a multicenter, randomized controlled, single-blind trial design. Based on the COVID-19 treatment regimen formulated by clinical guidelines, nebulized umbilical cord mesenchymal stem cell-derived exosomes (experimental group) or medically sterile saline solution (control group) will be administered to treat moderate, severe, and critically ill COVID-19 patients. By comparing the relief of symptoms and the occurrence of adverse events before and after treatment, the safety and effectiveness of umbilical cord mesenchymal stem cell-derived exosomes for the treatment of moderate, severe, and critically ill COVID-19 patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

(a) Voluntary participation of the patient and signing of the informed consent form; (b) The age of the patient at the time of signing the informed consent form should be ≥18 years old and ≤75 years old, regardless of gender; (c) The patient meets the criteria for moderate and severe patients with COVID-19 infection in China's "Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial Version 10)", as follows:

1. Moderate: continued fever >3 days and/or cough, dyspnea, or other symptoms, but respiratory rate (RR) <30 breaths/min, and oxygen saturation (SpO2) >93% at rest when inhaling air. Characteristic imaging manifestations of COVID-19 pneumonia can be observed (imaging is optional and can be included or excluded).
2. Severe: Any one of the following in adults cannot be explained by causes other than COVID-19 infection:

   1. dyspnea with RR ≥30 breaths/min.
   2. SpO2≤93% at rest when inhaling air.
   3. Ratio of partial pressure of arterial oxygen to fraction of inspired oxygen (PaO2/FiO2) ≤300 mmHg.
   4. Disease progression with significant increase in pulmonary lesions within 24-48 hours.
3. Critical: Any one of the following conditions:

   1. respiratory failure requiring mechanical ventilation.
   2. shock.
   3. other organ dysfunction requiring ICU monitoring and treatment. (d) Positive nucleic acid or antigen test; (e) No prior treatment with umbilical cord mesenchymal stem cell-derived exosomes; (f) The patient has a full understanding of the purpose and requirements of this trial and is willing to complete all trial procedures according to the trial requirements.

Exclusion Criteria:

(a) Female patients of childbearing age who are pregnant, lactating, or planning to conceive within the past year; (b) Severe heart, brain, kidney, hematopoietic system diseases, or other serious illnesses; (c) Neuro-muscular diseases causing impaired natural ventilation, including but not limited to spinal cord injury above the level of C5, amyotrophic lateral sclerosis, Guillain-Barre syndrome, and myasthenia gravis; (d) Currently undergoing hemodialysis or peritoneal dialysis; (e) Acute myocardial infarction within 30 days prior to screening; (f) Patients with lung or bone marrow transplantation; (g) History of epilepsy requiring continuous anticonvulsant treatment, or received anticonvulsant treatment within the past 3 years; (h) Active immunosuppression, defined as receiving immunosuppressive drugs or having medical conditions related to immunodeficiency. This includes:

1. HIV (AIDS or CD4<200 cells/mm3).
2. chemotherapy within 4 weeks before randomization.
3. long-term immunosuppressive therapy, including maintenance prednisone therapy (>40mg/day or equivalent for >1 month).
4. absolute neutrophil count <500/mm3. Exceptions are patients who have received short-term systemic (intravenous or oral) steroid treatment for <1 week or topical steroid treatment for skin disorders; (i) Patients with severe allergic reactions or contraindications to the treatment regimen in this study; (j) Patients with doubts about the treatment plan or obvious mental and psychological disorders; (k) Patients whom the investigator considers unsuitable for participation in this trial (such as factors that may reduce compliance with follow-up or refusal to accept relevant supportive treatment by the patient).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-01-23 (Estimated); Study Completion 2025-01-23 (Estimated)

PRIMARY OUTCOMES:
Symptom remission time after atomizing medication; | 3 months
  Symptom remission time after atomizing medication;
Improvement of serum inflammatory markers; | 3 months
  Improvement of serum inflammatory markers;
If there is baseline CT, CT review and comparison; | 3 months
  If there is baseline CT, CT review and comparison;

SECONDARY OUTCOMES:
Length of be hospitalized; | 3 months
  Length of be hospitalized;
Recovery time (nucleic acid turned negative) | 3 months
  Recovery time (nucleic acid turned negative)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Huang, Docter, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Background] El-Shennawy L, Hoffmann AD, Dashzeveg NK, McAndrews KM, Mehl PJ, Cornish D, Yu Z, Tokars VL, Nicolaescu V, Tomatsidou A, Mao C, Felicelli CJ, Tsai CF, Ostiguin C, Jia Y, Li L, Furlong K, Wysocki J, Luo X, Ruivo CF, Batlle D, Hope TJ, Shen Y, Chae YK, Zhang H, LeBleu VS, Shi T, Swaminathan S, Luo Y, Missiakas D, Randall GC, Demonbreun AR, Ison MG, Kalluri R, Fang D, Liu H. Circulating ACE2-expressing extracellular vesicles block broad strains of SARS-CoV-2. Nat Commun. 2022 Jan 20;13(1):405. doi: 10.1038/s41467-021-27893-2. PMID 35058437
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Yildirim F, Karaman I, Kaya A. Current situation in ARDS in the light of recent studies: Classification, epidemiology and pharmacotherapeutics. Tuberk Toraks. 2021 Dec;69(4):535-546. doi: 10.5578/tt.20219611. PMID 34957747
- [Background] Banerjee A, Pasea L, Harris S, Gonzalez-Izquierdo A, Torralbo A, Shallcross L, Noursadeghi M, Pillay D, Sebire N, Holmes C, Pagel C, Wong WK, Langenberg C, Williams B, Denaxas S, Hemingway H. Estimating excess 1-year mortality associated with the COVID-19 pandemic according to underlying conditions and age: a population-based cohort study. Lancet. 2020 May 30;395(10238):1715-1725. doi: 10.1016/S0140-6736(20)30854-0. Epub 2020 May 12. PMID 32405103
- [Background] Rubin R. Global Effort to Collect Data on Ventilated Patients With COVID-19. JAMA. 2020 Jun 9;323(22):2233-2234. doi: 10.1001/jama.2020.8341. No abstract available. PMID 32401275
- [Background] Liang W, Liang H, Ou L, Chen B, Chen A, Li C, Li Y, Guan W, Sang L, Lu J, Xu Y, Chen G, Guo H, Guo J, Chen Z, Zhao Y, Li S, Zhang N, Zhong N, He J; China Medical Treatment Expert Group for COVID-19. Development and Validation of a Clinical Risk Score to Predict the Occurrence of Critical Illness in Hospitalized Patients With COVID-19. JAMA Intern Med. 2020 Aug 1;180(8):1081-1089. doi: 10.1001/jamainternmed.2020.2033. PMID 32396163
- [Background] Wichmann D, Sperhake JP, Lutgehetmann M, Steurer S, Edler C, Heinemann A, Heinrich F, Mushumba H, Kniep I, Schroder AS, Burdelski C, de Heer G, Nierhaus A, Frings D, Pfefferle S, Becker H, Bredereke-Wiedling H, de Weerth A, Paschen HR, Sheikhzadeh-Eggers S, Stang A, Schmiedel S, Bokemeyer C, Addo MM, Aepfelbacher M, Puschel K, Kluge S. Autopsy Findings and Venous Thromboembolism in Patients With COVID-19: A Prospective Cohort Study. Ann Intern Med. 2020 Aug 18;173(4):268-277. doi: 10.7326/M20-2003. Epub 2020 May 6. PMID 32374815
- [Background] Carrade Holt DD, Wood JA, Granick JL, Walker NJ, Clark KC, Borjesson DL. Equine mesenchymal stem cells inhibit T cell proliferation through different mechanisms depending on tissue source. Stem Cells Dev. 2014 Jun 1;23(11):1258-65. doi: 10.1089/scd.2013.0537. Epub 2014 Mar 4. PMID 24438346
- [Background] Sauler M, Bazan IS, Lee PJ. Cell Death in the Lung: The Apoptosis-Necroptosis Axis. Annu Rev Physiol. 2019 Feb 10;81:375-402. doi: 10.1146/annurev-physiol-020518-114320. Epub 2018 Nov 28. PMID 30485762
- [Background] Naji A, Suganuma N, Espagnolle N, Yagyu KI, Baba N, Sensebe L, Deschaseaux F. Rationale for Determining the Functional Potency of Mesenchymal Stem Cells in Preventing Regulated Cell Death for Therapeutic Use. Stem Cells Transl Med. 2017 Mar;6(3):713-719. doi: 10.5966/sctm.2016-0289. Epub 2016 Oct 11. PMID 28297565
- [Background] Janockova J, Slovinska L, Harvanova D, Spakova T, Rosocha J. New therapeutic approaches of mesenchymal stem cells-derived exosomes. J Biomed Sci. 2021 May 25;28(1):39. doi: 10.1186/s12929-021-00736-4. PMID 34030679
- [Background] Yao J, Huang K, Zhu D, Chen T, Jiang Y, Zhang J, Mi L, Xuan H, Hu S, Li J, Zhou Y, Cheng K. A Minimally Invasive Exosome Spray Repairs Heart after Myocardial Infarction. ACS Nano. 2021 Jul 27;15(7):11099-11111. doi: 10.1021/acsnano.1c00628. Epub 2021 Jun 21. PMID 34152126
- [Background] Noori L, Arabzadeh S, Mohamadi Y, Mojaverrostami S, Mokhtari T, Akbari M, Hassanzadeh G. Intrathecal administration of the extracellular vesicles derived from human Wharton's jelly stem cells inhibit inflammation and attenuate the activity of inflammasome complexes after spinal cord injury in rats. Neurosci Res. 2021 Sep;170:87-98. doi: 10.1016/j.neures.2020.07.011. Epub 2020 Jul 25. PMID 32717259
- [Background] Park J, Kim S, Lim H, Liu A, Hu S, Lee J, Zhuo H, Hao Q, Matthay MA, Lee JW. Therapeutic effects of human mesenchymal stem cell microvesicles in an ex vivo perfused human lung injured with severe E. coli pneumonia. Thorax. 2019 Jan;74(1):43-50. doi: 10.1136/thoraxjnl-2018-211576. Epub 2018 Aug 3. PMID 30076187
- [Background] Zhang Y, Chen J, Fu H, Kuang S, He F, Zhang M, Shen Z, Qin W, Lin Z, Huang S. Exosomes derived from 3D-cultured MSCs improve therapeutic effects in periodontitis and experimental colitis and restore the Th17 cell/Treg balance in inflamed periodontium. Int J Oral Sci. 2021 Dec 14;13(1):43. doi: 10.1038/s41368-021-00150-4. PMID 34907166
- [Background] Joo HS, Suh JH, Lee HJ, Bang ES, Lee JM. Current Knowledge and Future Perspectives on Mesenchymal Stem Cell-Derived Exosomes as a New Therapeutic Agent. Int J Mol Sci. 2020 Jan 22;21(3):727. doi: 10.3390/ijms21030727. PMID 31979113
- [Background] Modani S, Tomar D, Tangirala S, Sriram A, Mehra NK, Kumar R, Khatri DK, Singh PK. An updated review on exosomes: biosynthesis to clinical applications. J Drug Target. 2021 Nov;29(9):925-940. doi: 10.1080/1061186X.2021.1894436. Epub 2021 Mar 12. PMID 33709876
- [Background] Morrison TJ, Jackson MV, Cunningham EK, Kissenpfennig A, McAuley DF, O'Kane CM, Krasnodembskaya AD. Mesenchymal Stromal Cells Modulate Macrophages in Clinically Relevant Lung Injury Models by Extracellular Vesicle Mitochondrial Transfer. Am J Respir Crit Care Med. 2017 Nov 15;196(10):1275-1286. doi: 10.1164/rccm.201701-0170OC. PMID 28598224
- [Background] Wu P, Zhang B, Shi H, Qian H, Xu W. MSC-exosome: A novel cell-free therapy for cutaneous regeneration. Cytotherapy. 2018 Mar;20(3):291-301. doi: 10.1016/j.jcyt.2017.11.002. Epub 2018 Feb 9. PMID 29434006
- [Background] Chu M, Wang H, Bian L, Huang J, Wu D, Zhang R, Fei F, Chen Y, Xia J. Nebulization Therapy with Umbilical Cord Mesenchymal Stem Cell-Derived Exosomes for COVID-19 Pneumonia. Stem Cell Rev Rep. 2022 Aug;18(6):2152-2163. doi: 10.1007/s12015-022-10398-w. Epub 2022 Jun 4. PMID 35665467
- [Background] Meng F, Xu R, Wang S, Xu Z, Zhang C, Li Y, Yang T, Shi L, Fu J, Jiang T, Huang L, Zhao P, Yuan X, Fan X, Zhang JY, Song J, Zhang D, Jiao Y, Liu L, Zhou C, Maeurer M, Zumla A, Shi M, Wang FS. Human umbilical cord-derived mesenchymal stem cell therapy in patients with COVID-19: a phase 1 clinical trial. Signal Transduct Target Ther. 2020 Aug 27;5(1):172. doi: 10.1038/s41392-020-00286-5. PMID 32855385
- [Background] Song NJ, Allen C, Vilgelm AE, Riesenberg BP, Weller KP, Reynolds K, Chakravarthy KB, Kumar A, Khatiwada A, Sun Z, Ma A, Chang Y, Yusuf M, Li A, Zeng C, Evans JP, Bucci D, Gunasena M, Xu M, Liyanage NPM, Bolyard C, Velegraki M, Liu SL, Ma Q, Devenport M, Liu Y, Zheng P, Malvestutto CD, Chung D, Li Z. Treatment with soluble CD24 attenuates COVID-19-associated systemic immunopathology. J Hematol Oncol. 2022 Jan 10;15(1):5. doi: 10.1186/s13045-021-01222-y. PMID 35012610